CLINICAL TRIAL: NCT06346678
Title: Accuracy of Accuhaler Tester, Ellipta Tester and Turbutester in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Narongkorn Saiphoklang, MD, Associate Professor, Thammasat University
Other Study IDs: MTU-EC-IM-0-016/67
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; COPD; Accuhaler tester; Ellipta tester; Turbutester; Peak inspiratory flow rate
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Accuhaler tester — Patients will perform testing with Accuhaler tester, Ellipta tester and Turbutester.
  Other Names: Ellipta tester; Turbutester

SUMMARY:
The goal of this observational study is to investigate the accuracy of Accuhaler tester, Ellipta tester and Turbutester in patients with chronic obstructive pulmonary disease (COPD). The main question it aims to answer is:

• Do Accuhaler tester, Ellipta tester, and Turbutester demonstrate comparable accuracy to the In-check DIAL for assessing inspiratory inhalation force in COPD patients?

DETAILED DESCRIPTION:
This study is a cross-sectional study. COPD patients aged 40 years or older will be included. Peak inspiratory flow rate (PIFR) will be assessed using In-check DIAL as the standard tool. PIFR will be tested in each patient using Accuhaler tester, Ellipta tester and Turbutester.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis with confirmed by post-bronchodilator forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) <0.7
* Age 40 years or older
* Smoking history 10 pack-years or more

Exclusion Criteria:

* COPD exacerbation within 3 months
* Oral or intravenous corticosteroid treatment within 6 weeks
* Inability to perform assessment of peak inspiratory flow rate
* Asthma
* Tracheostomy, invasive or noninvasive mechanical ventilation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients aged 40 years or older who are confirmed diagnosis by spirometry (post-bronchodilator FEV1/FVC <0.7) and smoking history 10 pack-years or more.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Accuracy of Accuhaler tester | At day 1 of the study
  Percentage
Accuracy of Ellipta tester | At day 1 of the study
  Percentage
Accuracy of Turbutester | At day 1 of the study
  Percentage

SECONDARY OUTCOMES:
Prevalence of suboptimal peak inspiratory flow rate | At day 1 of the study
  Percentage
Prevalence of insufficient peak inspiratory flow rate | At day 1 of the study
  Percentage

CONTACTS AND LOCATIONS:
Overall Officials: Narongkorn Saiphoklang, MD, Principal Investigator — Thammasat University Faculty of Medicine
Locations (1):
- Narongkorn Saiphoklang, Pathum Thani, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Yes
IPD and documents will be available for sharing immediately after publication for a period of 2 years.
Supporting Information: Study Protocol, SAP, CSR